CLINICAL TRIAL: NCT02956889
Title: A Single Arm, Phase II, Multicenter Study To Assess The Efficacy And Safety Of Vismodegib And Radiotherapy In Patients With High Risk Or Locally Advanced Basal Cell Carcinoma Not Amenable To Radical Surgery
Brief Title: To Assess The Efficacy And Safety Of Vismodegib And Radiotherapy In Advanced Basal Cell Carcinoma
Acronym: virgilio
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2015-001
Record Dates: First submitted 2016-07-20; First posted 2016-11-07 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Carcinoma, Basal Cell
Keywords: Carcinoma, Basal Cell; Vismodegib; Radiotherapy
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vismodegib & Radiotherapy (Experimental): Radiotherapy (RT) will be administered with a total dose of 50 Gy/2.5 Gy per fraction over 4 weeks.
  Treatment with Vismodegib will start within 4 weeks by the end of radiotherapy and will continue for 6 cycles
  Interventions: Drug: Vismodegib; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Vismodegib — Patients will receive a continuous once-daily oral dosing of Vismodegib at a dosage of 150 mg .
  Other Names: Erivedge
Radiation: Radiotherapy — Radiotherapy (RT) will be administered with a total dose of 50 Gy/2.5 Gy per fraction over 4 weeks.

SUMMARY:
This is a Fleming-A' Hern, single arm, multicenter, no-profit, phase II study of radiotherapy and Vismodegib in adult patients with high risk or locally advanced basal cell carcinoma not amenable to radical surgery cell carcinoma (BCC) (comparator: not applicable).

The recruitment period is expected to be approximately 24 months. The trial will consist of a Screening/Baseline period (Day -28 to -1), a Treatment Period when patients will be treated with radiotherapy (4 weeks) followed by Vismodegib 150 mg/die continuously for six cycles (24 weeks).

The study will end 14 months after start of treatment of the last patient enrolled and evaluable according to primary end point.

DETAILED DESCRIPTION:
This is a Fleming-A' Hern, single arm, multicenter, no-profit, phase II study of radiotherapy and Vismodegib in adult patients with high risk or locally advanced basal cell carcinoma not amenable to radical surgery cell carcinoma (BCC) (comparator: not applicable).

The recruitment period is expected to be approximately 24 months. The trial will consist of a Screening/Baseline period (Day -28 to -1), a Treatment Period when patients will be treated with radiotherapy (4 weeks) followed by Vismodegib 150 mg/die continuously for six cycles (24 weeks).

The study will end 14 months after start of treatment of the last patient enrolled and evaluable according to primary end point.

The primary objective is to evaluate the activity of the study therapy (radiotherapy followed by six cycles of Vismodegib 150 mg/d continuously) in terms of proportion of patients progression free at 12 months.

The secondary objectives are: to evaluate the efficacy of the study therapy in terms of progression free survival (PFS) and overall survival (OS); to assess the response in terms of overall response rate (ORR) (complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD)); to assess duration of response (DoR); to assess the safety in terms of incidence, type, and severity of adverse events (AEs) and serious adverse events (SAEs) ;to measure the effects of skin disease on quality of life (QoL) of patients under therapy (Skindex-16)

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed informed consent
2. Age ≥ 18 years
3. Histopathologic confirmation that the lesion is BCC before enrollment
4. Patients with high risk of relapse BCC not undergone radical surgery, for which treating physician must consider the disease to be no more operable.
5. Clinical features defining high risk of relapse include infiltrative growth margins, size, tumor location, histological subtype (the morpheaform, the sclerosing, the infiltrating, the micronodular and the metatypical subtypes are associated with higher risk of relapse as compared to the risk associated with the superficial and the nodular types), recurrent-refractory tumors (see Table 1), basal cell carcinoma size (largest tumor diameter) ≤ 5 cm for head and neck tumors
6. Clinical features for definition of "BCC not amenable for radical surgery" include:

   * BCC that has recurred in the same location after minimum 2 surgical procedures (excluding biopsies) and/or curative resection is deemed unlikely
   * multifocal BCC or extensive tumors (see table 1) with bleeding or infected areas
   * anticipated substantial morbidity and/or deformity from surgery (e.g., removal of all or part of a facial structure, such as nose, ear, eyelid, eye; or requirement for limb amputation)
7. Patients with BCCs localized where surgery is technically difficult, or would result in unacceptable tissue destruction
8. Patients with a clinical contraindication to surgery
9. Previous radiotherapy on other BCC
10. Patients with measurable and/or non-measurable disease (as defined by RECIST, v1.1) are allowed
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
12. Adequate hematopoietic capacity, defined as the following:

    * Hemoglobin : 8.5 g/dl
    * Absolute neutrophil count (ANC) ≥ 1500/mL
    * Platelet count ≥ 75,000/mL
13. Adequate hepatic function, defined as the following:

    Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN)Total bilirubin ≤ 1.5 × ULN or within 3 × ULN for patients with documented Gilbert syndrome. Adequate renal function, defined by calculated serum creatinine clearance (CrCl) ≥ 30 mL/min
14. For women of childbearing potential, a negative serum pregnancy test within 7days prior to commencement of dosing is required.
15. Women of child-bearing potential must use two methods of acceptable contraception including one highly effective method and a barrier method, as directed by their physician, during treatment and for at least 24 months after completion of study treatment. Highly effective methods of contraception are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (e.g., implants, injectables, combined oral contraception, or intra-uterine devices). At the discretion of the Investigator, acceptable methods of contraception may include total abstinence. Periodic abstinence (e.g., calendar, ovulation, symptothermal, and post ovulation methods) and withdrawal are not acceptable methods of contraception (See Appendix B).
16. For male patients with female partners of childbearing potential, agreement to use a condom, even after a vasectomy, during sexual intercourse with female partners while being treated with Vismodegib, and for 2 months after completion of study treatment
17. Agreement not to donate blood or blood products during the study and for at least 24 months after completion of study treatment (Vismodegib).

Exclusion Criteria:

1. Inability or unwillingness to swallow capsules
2. Inability or unwillingness to comply with study procedures
3. Pregnancy or lactation (lactation not allowed for at least 24 months after completion of study treatment)
4. Concurrent non-protocol-specified anti-tumor therapy (e.g., chemotherapy, other targeted therapy, photodynamic therapy, including participation in an experimental drug study)
5. Metastatic BCC
6. Gorlin Syndrome or any other contraindication to radiotherapy
7. Recent (i.e., within the past 28 days prior to enrollment in this study) or current participation in another experimental drug study
8. Uncontrolled medical illness, including advanced malignancies, at the discretion of the Investigator
9. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
evaluate the activity of the study therapy in terms of proportion of patients progression free | 1 years
  The primary objective is to evaluate the activity of the study therapy (radiotherapy followed by six cycles of Vismodegib 150 mg/d continuously) in terms of proportion of patients progression free at 12 months.

SECONDARY OUTCOMES:
evaluate the efficacy of the study therapy in terms of progression free survival | 2 years
  The secondary objectives are: to evaluate the efficacy of the study therapy in terms of progression free survival (PFS)
evaluate the efficacy of the study therapy in terms overall survival | 2 years
  The secondary objectives are: to evaluate the efficacy of the study therapy in terms of overall survival (OS);
response in terms of overall response rate (ORR) | 2 years
  to assess the response in terms of ORR (complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD))
duration of response | 2 years
  to assess duration of response (DoR);
assess the safety in terms of incidence, type, and severity of adverse events (AEs) and serious adverse events (SAEs) | 2 years
  to assess the safety in terms of incidence, type, and severity of AEs and SAEs
measure the effects of skin disease on quality of life (QoL) of patients | 2 years
  to measure the effects of skin disease on quality of life (QoL) of patients under therapy (Skindex-16)

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico humanitas, Rozzano, Mi, Italy

IPD SHARING:
Plan to Share IPD: No
not planned

REFERENCES:
- [Background] Diffey BL, Langtry JA. Skin cancer incidence and the ageing population. Br J Dermatol. 2005 Sep;153(3):679-80. doi: 10.1111/j.1365-2133.2005.06799.x. No abstract available. PMID 16120172
- [Background] Gailani MR, Stahle-Backdahl M, Leffell DJ, Glynn M, Zaphiropoulos PG, Pressman C, Unden AB, Dean M, Brash DE, Bale AE, Toftgard R. The role of the human homologue of Drosophila patched in sporadic basal cell carcinomas. Nat Genet. 1996 Sep;14(1):78-81. doi: 10.1038/ng0996-78. PMID 8782823
- [Background] Von Hoff DD, LoRusso PM, Rudin CM, Reddy JC, Yauch RL, Tibes R, Weiss GJ, Borad MJ, Hann CL, Brahmer JR, Mackey HM, Lum BL, Darbonne WC, Marsters JC Jr, de Sauvage FJ, Low JA. Inhibition of the hedgehog pathway in advanced basal-cell carcinoma. N Engl J Med. 2009 Sep 17;361(12):1164-72. doi: 10.1056/NEJMoa0905360. Epub 2009 Sep 2. PMID 19726763
- [Background] Telfer NR, Colver GB, Morton CA; British Association of Dermatologists. Guidelines for the management of basal cell carcinoma. Br J Dermatol. 2008 Jul;159(1):35-48. doi: 10.1111/j.1365-2133.2008.08666.x. PMID 18593385
- [Background] Sekulic A, Migden MR, Oro AE, Dirix L, Lewis KD, Hainsworth JD, Solomon JA, Yoo S, Arron ST, Friedlander PA, Marmur E, Rudin CM, Chang AL, Low JA, Mackey HM, Yauch RL, Graham RA, Reddy JC, Hauschild A. Efficacy and safety of vismodegib in advanced basal-cell carcinoma. N Engl J Med. 2012 Jun 7;366(23):2171-9. doi: 10.1056/NEJMoa1113713. PMID 22670903
- [Background] Chang AL, Solomon JA, Hainsworth JD, Goldberg L, McKenna E, Day BM, Chen DM, Weiss GJ. Expanded access study of patients with advanced basal cell carcinoma treated with the Hedgehog pathway inhibitor, vismodegib. J Am Acad Dermatol. 2014 Jan;70(1):60-9. doi: 10.1016/j.jaad.2013.09.012. Epub 2013 Nov 1. PMID 24189279
- [Background] Tang JY, Mackay-Wiggan JM, Aszterbaum M, Yauch RL, Lindgren J, Chang K, Coppola C, Chanana AM, Marji J, Bickers DR, Epstein EH Jr. Inhibiting the hedgehog pathway in patients with the basal-cell nevus syndrome. N Engl J Med. 2012 Jun 7;366(23):2180-8. doi: 10.1056/NEJMoa1113538. PMID 22670904
- [Background] Strasswimmer JM. Potential Synergy of Radiation Therapy With Vismodegib for Basal Cell Carcinoma. JAMA Dermatol. 2015 Sep;151(9):925-6. doi: 10.1001/jamadermatol.2015.0977. No abstract available. PMID 25874820
- [Background] Pollom EL, Bui TT, Chang AL, Colevas AD, Hara WY. Concurrent Vismodegib and Radiotherapy for Recurrent, Advanced Basal Cell Carcinoma. JAMA Dermatol. 2015 Sep;151(9):998-1001. doi: 10.1001/jamadermatol.2015.0326. PMID 25874733